CLINICAL TRIAL: NCT02874053
Title: The Role of Emotions and Regulatory Focus in Decision Making That Involves Risk Tradeoffs
Status: Withdrawn | Type: Observational
Why Stopped: PI left the NIH
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916161; 16-C-N161
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: Risk Perceptions; Medical Tradeoffs; Regulatory Focus; Integral Affect
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Healthy: Healthy Volunteers

SUMMARY:
Background:

People with cancer often have to make complex decisions about their treatment. For some of these decisions, they have to weigh the benefits of a treatment against its side effects. They may have to think about its potential to increase the risk of another disease. One example is hormone replacement therapy. That reduces a woman s risk of getting colorectal cancer, but it raises her risk of getting breast cancer. Researchers want to learn more about how people make tradeoff decisions like these.

Objective:

To learn about how people respond to information about hypothetical health and medical treatment options.

Eligibility:

Adults ages 18 70.

Design:

Participants will have one 30-minute visit.

Participants will complete a series of short questionnaires. These will be about their beliefs and values. Some may be about cancer and heart disease risk. Participants ages 18 to 29 will answer questions about sexual health.

Participants will write a paragraph or two about a room in their house or about a life event.

Participants will read a series of stories. These will describe different hypothetical health treatments.

The stories describe a pill that lowers the risk of one health condition, but raises the risk for another. After each story, participants will note how willing they are to take the pill.

Participants will answer questions about the information that they got. They will also answer questions about their health, beliefs, and opinions.

Participants will do 2 attention tasks computer.

DETAILED DESCRIPTION:
Given that many preventive and therapeutic treatments for cancer lower the risk of one disease, but increase the risk of another disease (or have substantial side effects), patients and doctors often must make medical decisions that involve tradeoffs. When faced with these tradeoffs, people make decisions based on factors beyond objective probability estimates. Emotions and regulatory focus are known to influence judgment and risk propensity in non-tradeoff decision-making contexts, but little is known about their independent and joint effects on decision making in tradeoff scenarios where both options involve some degree of risk. This study aims to generate fundamental knowledge about how individuals make decisions in the context of these tradeoffs, and whether individuals with clinical disorders or at risk for clinical disorders differ from healthy individuals in their decision making. This will have immediate translational potential for applied studies of decision making among cancer patients and those at increased risk for cancer. We plan to examine the effects of discrete incidental affect on tradeoff decision making, and the role of regulatory focus as a moderator of its effect. During visits to a laboratory at the University of Pittsburgh, human subjects aged 18 to 70 will be randomly assigned to write about an emotional event (something that made them angry or afraid depending on study condition) or about a room in their house (neutral emotion condition). Then, they will read a series of scenarios that describe a pill that lowers their risk of one health condition, but raises their risk for another. After each, they will indicate their willingness to take the pill. Regulatory focus, risk perceptions, and implicit measures of risk propensity and anticipated emotions will also be assessed. Drawing on previous research, we hypothesize that participants asked to recall an angry experience will be more willing to take the pill, and that this effect will be particularly strong for those with a promotion-oriented regulatory focus. Prevention-focused participants asked to recall an experience that made them feel afraid are expected to be least willing to take the pill. We will also explore possible mechanisms underlying the emotion induction s effect on pill choice, such as shifts in risk perceptions, biased attentional focus, and implicitly measured anticipated emotions.

ELIGIBILITY:
* INCLUSION CRITERIA:

For Study A, community members will be invited to participate if they are aged 18 to 70.

For Study B, University at Pittsburgh students will be invited to participate if they are aged 18 and over.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community members and students from the University of Pittsburgh.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
willingness to take hypothetical pill | at baseline (cross-sectional)
  self-reported behavioral willingness

CONTACTS AND LOCATIONS:
Overall Officials: William M Klein, Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Lockwood P, Jordan CH, Kunda Z. Motivation by positive or negative role models: regulatory focus determines who will best inspire us. J Pers Soc Psychol. 2002 Oct;83(4):854-64. PMID 12374440
- [Background] Waters EA, Weinstein ND, Colditz GA, Emmons KM. Aversion to side effects in preventive medical treatment decisions. Br J Health Psychol. 2007 Sep;12(Pt 3):383-401. doi: 10.1348/135910706X115209. PMID 17640453